CLINICAL TRIAL: NCT02180815
Title: ReVENT Sleep Apnea System, a Minimally Invasive Approach to Treat Obstructive Sleep Apnea: a Prospective Multicenter Post-Market Observational Study
Brief Title: REV 002 Observational Study of the ReVENT Sleep Apnea System: Minimally Invasive Treatment for Obstructive Sleep Apnea
Status: Terminated | Type: Observational
Why Stopped: Sufficient follow-up information obtained to support study goals
Sponsor: Revent Medical International B.V. (Industry)
Collaborators: Revent Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: REV 002
Record Dates: First submitted 2014-06-11; First posted 2014-07-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Obstructive Sleep Apnea due to primary tongue base closure; Minimally invasive surgery; ReVENT Sleep Apnea System; Tongue implants
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ReVENT implanted group
  Interventions: Device: ReVENT Sleep Apnea System

INTERVENTIONS:
Device: ReVENT Sleep Apnea System

SUMMARY:
The purpose of this post-market observational study is to assess the effectiveness and patient perception of benefit of the ReVENT Sleep Apnea System in patients diagnosed with Obstructive Sleep Apnea due to primary tongue base closure. The ReVENT Sleep Apnea System is a minimally invasive surgical approach to treat Obstructive Sleep Apnea. The ReVENT Sleep Apnea System consists of an implanter kit and tongue implants. The implants are permanently implanted in the tongue during a minimally invasive outpatient surgical procedure to prevent tongue base closure during sleep.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Obstructive Sleep Apnea due to primary tongue base closure.
* AHI ≥ 10 and AHI ≤ 40 (at least 90% of apneas and hypopneas must be obstructive).
* BMI ≤ 32.
* Confirmation of tongue base closure as the primary source of obstruction with Drug Induced Sleep Endoscopy (DISE).

Exclusion Criteria:

* Patient with prior tongue-base surgery
* Uvulopalatopharyngoplasty, soft palate surgery, tonsillectomy or minimally invasive RF ablation of the tongue within the last six (6) months.
* History of mandibular and/or hyoid advancement to treat OSA.
* Any contraindications as listed in the approved Instructions for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Obstructive Sleep Apnea due to primary tongue base closure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in Apnea-Hypopnea Index (AHI) | 3, 6 and 12 months

SECONDARY OUTCOMES:
Patient perception of benefit as measured by change in daytime sleepiness and sleep-related quality of life | 3, 6 and 12 months

OTHER OUTCOMES:
Safety profile assessed by incidence of adverse events | 1 week, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Wolfgang Bergler, Principal Investigator — St. Joseph-Stift
Locations (14):
- Belgium (2):
  - Cliniques Universitaires Saint Luc, Brussels
  - University Hospital Antwerp, Edegem
- Pavelec LENTE, Ltd., Pilsen, Czechia
- Germany (7):
  - St Joseph-Stift, Bremen
  - St. Franziskus Hospital HNO-Klinik, Cologne
  - Alfried Krupp Krankenhaus, Essen
  - Asklepios Klinik Harburg, Hamburg
  - Universitäts-HNO-Klinik Mannheim, Mannheim
  - Klinikum Ernst von Bergmann, Potsdam
  - Universitätsklinikum HNO-Klinik, Ulm
- Netherlands (3):
  - MC Slotervaart, Amsterdam
  - Sint Antonius Hospital, Nieuwegein
  - ISALA Afdeling KNO-Heelkunde Isala, Zwolle
- Cantonal Hospital Baselland - ENT Department, Liestal, Switzerland